CLINICAL TRIAL: NCT02503384
Title: Clinical and Basic Study for Pediatric Liver Transplantation
Acronym: CBSPLT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 15411950401
Record Dates: First submitted 2015-07-17; First posted 2015-07-21 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Biliary Atresia; Metabolic Disorders; Fulminant Liver Failure; Hepatic Tumors
MeSH Terms: conditions — Biliary Atresia; Metabolic Diseases; Liver Failure, Acute; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Background: In mainland China, the development of pediatric liver transplantation (LT) has lagged behind that of adult LT during the past two decades, but it has been progressing immensely in recent years. Renji hospital(shanghai) is currently the largest pediatric transplant center in mainland China.

Aim and method: This study is performed for establishment of key techniques for pediatric LT in mainland China, including the indications and timing for pediatric LT, the criteria for donor selections, living donor LT planning, prevention and treatment for posttransplant complications, long-term follow-up management et al.

DETAILED DESCRIPTION:
Outcome measures:

* Annual caseloads of pediatric liver transplantation
* Patient survival: 1-, 3- and 5-year patient survival after liver transplantation
* Graft survival: 1-, 3- and 5-year graft survival after liver transplantation
* Posttransplant complications, such as biliary complications, vascular complications, acute rejections, infections et al.
* Perioperative data, such as duration of operations, postoperative hospital stay et al.
* Clinical data for living donors.

ELIGIBILITY:
Inclusion Criteria:

* Children with end-stage liver diseases
* Children with metabolic disorders for whom liver transplantation are required
* Children with fulminant liver failure
* Children with unresectable hepatic tumors
* Other miscellaneous conditions which need liver transplantation

Exclusion Criteria:

* Recipient age ≥ 18 years
* Patients with metastatic liver tumors
* Severe systmatic infections
* Acquired Immune Deficiency Syndrome

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric liver transplantation cases
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-07 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Patient survival | up to 36 months
Graft survival | up to 36 months
Annual caseload for pediatric liver transplantation | up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Xia, MD, PhD, Study Chair — Department of Liver Surgery, Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Deparment of Liver Surgery, Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, China